CLINICAL TRIAL: NCT00174850
Title: A 14 Week Open-Label Study to Evaluate the Tolerability of Switching From an SSRI to Tiagabine(GABITRIL) in Order to Alleviate SSRI Induced Sexual Dysfunction in Generalized Anxiety Disorder Patients
Brief Title: Switching From an SSRI to Tiagabine(GABITRIL) in Order to Alleviate SSRI Induced Sexual Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4984; 1042242-1; 33625
Record Dates: First submitted 2005-09-14; First posted 2005-09-15 (Estimated); Last update posted 2008-09-18 (Estimated); Status verified 2008-09

CONDITIONS: Anxiety; Sexual Dysfunction
Keywords: anxiety; sexual dysfunction; ssri
MeSH Terms: conditions — Anxiety Disorders; Sexual Dysfunction, Physiological

INTERVENTIONS:
Drug: Gaitril

SUMMARY:
Anxious patients are now treated with Selective Serotonin Reuptake Inhibitor medications (common antidepressants) which elevate serotonin and thus alleviate anxiety. These medications have clearly proven efficacy upwards of 70% for many anxiety disorders. In regards to tolerability, they have a major problem in that they often produce sexual dysfunction in men and women (ie. decreased libido, anorgasmia, impotence) upwards of 30% of the time.

Benzodiazepine anxiolytics are also FDA approved to treat anxiety with equal efficacy and greater tolerability (very little, if any sexual dysfunction). They do, however, carry a substantial risk for addiction. Tiagabine is a Selective GABA Reuptake Inhibitor (SGRI) that is FDA approved to treat certain types of epilepsy. Like benzodiazepines, Tiagabine also increases the neurotransmitter, GABA, in the brain and is thought to alleviate anxiety (see references below) this way too, but without any addiction risk common to Valium-type drugs. The safety profile of Tiagabine is thought to be much safer. Two double blind studies are ongoing which are looking at Tiagabine's effectiveness in PTSD and GAD. There are many open label studies showing anxiety reduction and many psychiatrists in clinical practice are utilizing this agent as an anxiety treatment in an off-label manner.

This study is designed to evaluate anxious patients who are taking SSRI medication, have had a reasonable response, but are experiencing significant sexual side effects which are pushing them towards noncompliance and possible relapse into anxiety. 30 subjects (15 men and 15 women) will be asked to join the study and be placed on Tiagabine as well as their current SSRI. Once an acceptable dose of Tiagabine is reached in the first four weeks, the subjects' SSRIs will be slowly stopped. Two weeks after enrollment, all subjects will be called in order to check for any side effects to the study drug and to insure that each subject is titrating to the proper dose of study drug according to the study protocol. An open-label, non-placebo prospective 10 week follow up will occur, where the now Tiagabine monotherapy subjects will be followed to see primarily if their sexual dysfunction improves and if there anxiety remains controlled.

DETAILED DESCRIPTION:
This is an open-label (no placebo) study to see if a change from SSRI to Tiagabine may alleviate sexual dysfunction while maintaining subject in a non-anxious state. 30 Subjects ( at least 50% female) will currently be taking a single SSRI for at least 4 weeks and report at least a 50% drop in their anxiety severity as a result. They must also report a chronological emergence of sexual dysfunction ( decreased sex drive, arousal, lubrication, or onset of impotence, anorgasmia or delayed ejaculation) following the SSRI initiation.

Subjects will complete consenting process and attend a screening visit where they will be given a MINI psychiatric diagnostic evaluation to confirm anxiety disorder, be given a Hamilton Anxiety and a Hospital Anxiety & Depression Scale evaluation to delineate current anxiety level (secondary measure). They will also complete self rated sexual health scales such as the ASEX to assess sexual functioning (primary measure). Subjects will undergo a brief physical exam and bloodwork will be ordered if the patient has an underlying medical condition that warrants this type of medical clearance. The same would hold true if an EKG is needed. Neither SSRIs, nor tiagabine warrants blood monitoring or EKGs per the FDA.

Assuming subject meets eligibility, they will start titrating upwards as tolerated on tiagabine and downwards on their SSRI. Titration with Tiagabine is flexible but typically starts at the night of Day 1: 4 mg/day (2mg qAm with breakfast and 2mq qHS before bedtime with a snack for five days). On day 6: 8mg/day (2mg with breakfast and 6mg before bedtime with a snack). Day 13: 12mg/day in split doses: (4mg am with breakfast and 8mg before bedtime with a snack). Two weeks after enrollment, all subjects will be called in order to check for any side effects to the study drug and to insure that each subject is titrating to the proper dose of study drug according to the study protocol. At the discretion of the investigator, dosing may be lowered to alleviate side effects. Vist 2 will occur at the end of week 4 when all SSRI is off and optimal tiagabine is in place. All scales except MINI will be completed. Vist 3 will occur at the end of week 8 and scales will be completed. Visit 4 will be the final visit at end of week 14, scales, PE and blood/EKG collected as warranted. The efficacy and safety of Tiagabine will be evaluated throughout the treatment period (see flow chart). At the end of the study, subjects may opt to continue tiagabine or be titrated back to their SSRI. Our team will also liaison with the subject's prescriber to ensure follow up and continuity of care after study exit.

ELIGIBILITY:
Inclusion Criteria: Patients are included in the study if all of the following criteria are met:

1. Written informed consent is obtained.
2. The patient is English-speaking and 18 through 64 years of age inclusive.
3. The patient meets the DSM-IV criteria for generalized anxiety disorder as determined by the MINI and psychiatric evaluation.
4. The patient is currently responding to and taking a monotherapy SSRI (including venlafaxine) for ≥ 4 weeks and on a stable, adequate therapeutic for ≥ 4 weeks
5. the patient reports clear sexual side effects post dating the SSRI start
6. The patient has a total score of at less than 18 on the HAM-A scale

(i) The patient is in good health as determined by a medical and psychiatric history, medical examination, (j) Women must be of nonchildbearing potential [i.e., postmenopausal, be surgically sterile (hysterectomy or tubal ligation)] or must meet all of the following conditions: using a reliable, medically accepted form of contraception for at least 60 days before the baseline visit, and agree to continue such use throughout the duration of the study and for 30 days after the final dose of study drug. Reliable forms of contraception include oral, implanted, or injected contraceptives; intrauterine devices in place for at least 3 months; and adequate barrier methods in conjunction with spermicide (abstinence is considered an acceptable contraceptive regimen). Women must be given a pregnancy test (ßHCG), unless they are at least 2 years postmenopausal or surgically sterile, and the results of the test must be negative.

(k) The patient must be willing and able to comply with study restrictions and to remain at the clinic for the required duration during the study period, and willing to return to the clinic for the follow-up evaluation as specified in this protocol.

Exclusion Criteria: Patients are excluded from participating in this study if 1 or more of the following criteria are met:

1. Other current mental illness/disorder
2. The patient is a significant risk of suicide

(d) The patient has a history of greater than one previous depressive episode or has not been in remission >1 year (e) The patient cannot take sildenafil or any other sexually enhancing agent (f) The patient has any serious, unresolved or unstable medical and/or psychiatric condition (treated or untreated).

(g) The patient has previously participated in any clinical study with GABITRIL or treated with GABITRIL.

(h) The patient is a pregnant or lactating woman (women becoming pregnant during the study will be withdrawn from the study).

(l) The patient has used an investigational drug within 1 month before the screening visit or is participating in a concurrent clinical trial.

(m) The patient has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including gastrointestinal surgery) or have an explainable medical condition causing sexual dysfunction (n) The patient has had alcohol or sedative dependence within last one year or any other illegal substance abuse/dependence in last 3 months including heavy caffeine, nicotine use contributing to anxiety state (o) The patient is unlikely to comply with the study protocol, be unreliable in providing ratings, or is unsuitable for any reason, as judged by the investigator.

(p) The patient has a clinically significant deviation from normal in the physical examination.

-

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30
Dates: Start 2004-07; Study Completion 2005-05

PRIMARY OUTCOMES:
none as yet, date being analyzed

SECONDARY OUTCOMES:
none as yet.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L. Schwartz, MD, Principal Investigator — SUNY Upstate Medical University, Psychiatry Dept.
Locations (1):
- Psychiatry Dept. SUNY Upstate Medical University, Syracuse, New York, United States